CLINICAL TRIAL: NCT02551172
Title: An Efficacy and Safety Study of HCP1105 Capsule in Combined Hyperlipidemic Patients With High Risk for Coronary Heart Disease (CHD): A Randomized,Double-blind, Multicenter, Phase 3 Study
Brief Title: Evaluating the Efficacy and Safety of HCP1105 in Combined Hyperlipidemic Patients With High Risk for CHD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ROMA-301
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental sequence (Experimental): Run-in period → Treatment period HGP0816 20mg 1tab HCP1105 4capsues +Placebo of HGP0816
  Interventions: Drug: HCP1105; Drug: HGP0816; Drug: Placebo of HGP0816
- comparative sequence (Placebo Comparator): Run-in period → Treatment period HGP0816 20mg 1tab Placebo of HCP1105 4capsues +HGP0816 20mg
  Interventions: Drug: HGP0816; Drug: Placebo of HCP1105

INTERVENTIONS:
Drug: HCP1105 — Rosuvastatin + Omega-3-acids ethyl esters
  Arms: experimental sequence
Drug: HGP0816 — Rosuvastatin
Drug: Placebo of HCP1105 — Soybean Oil
  Arms: comparative sequence
Drug: Placebo of HGP0816 — Exclusion of Rosuvastatin in HGP0816
  Arms: experimental sequence

SUMMARY:
To investigate the efficacy and safety after administration of HCP1105 in hyperlipidemic patients with high risk for CHD.

DETAILED DESCRIPTION:
An efficacy and safety study of HCP1105 Capsule in combined hyperlipidemic patients with high risk for Coronary Heart Disease(CHD): A randomized,double-blind, multicenter, phase 3 study.

ELIGIBILITY:
Inclusion Criteria:

* age 19≤
* Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

* History of clinically significant hypersensitivity reaction with HMG-CoA reductase inhibitor and Omega-3
* Subject who has active liver disease and severe liver failure(Continuous elevation of AST,ALT level with unspecified cause or AST, ALT level exceeds more than three times of maximum upper range.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Mean rate of change of non-HDL-C (%) from baseline | 12 weeks

SECONDARY OUTCOMES:
Mean rate of change of HDL-C (%) from baseline | 4, 8, 12 weeks
Mean rate of change of LDL-C (%) from baseline | 4, 8, 12 weeks
Mean rate of change of Triglyceride (%) from baseline | 4, 8, 12 weeks
Mean rate of change of Total cholesterol (%) from baseline | 4, 8, 12 weeks
Mean rate of change of Total apo A1 (%) from baseline | 4, 8, 12 weeks
Mean rate of change of Total apo B (%) from baseline | 4, 8, 12 weeks
Mean rate of change of Lipoprotein(a) (%) from baseline | 4, 8, 12 weeks
Mean rate of change of hs-CRP (%) from baseline | 4, 8, 12 weeks
Rate of the subjects who meet the target level of treatment | 4, 8, 12 weeks
  target level (Non-HDL-C<130mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-yeol Park, M.D., Ph.D., Principal Investigator — Asan Medecal Center
Locations (1):
- Euljii General Hospital, Seoul, Seoul, South Korea